CLINICAL TRIAL: NCT03028792
Title: Attention Training for Underserved Youth With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Susanna Chang, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#15-000334
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Anxiety
Keywords: attention training, youth, latino
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Modification Training (Experimental): Attention Modification Program Active computer-based attention training treatment designed to directly but implicitly modify biased attention patterns in anxious patients in service of symptom relief. AMP is a modified version of the dot-probe paradigm similar to the original task used by MacLeod, Mathews, and Tata. This paradigm has been modified to facilitate an attention bias away from threatening material. In this case, the probe always replaces the neutral stimuli.
  Interventions: Behavioral: Attention Modification Program
- Attention Control Training (Sham Comparator): Placebo Comparator: Attention Control Condition Control computer-based attention training task, which is not designed to modify biased attention patterns in anxious patients. ACC is a modified version of the dot-probe paradigm similar to the original task used by MacLeod, Mathews, and Tata. In this case, the probe randomly replaces the neutral stimuli or the threat stimuli.
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: Attention Modification Program — Each trial begins with a fixation cross at the center of the computer screen for 500 ms. The cross is then replaced by a face pair presented in the center of the screen. The face pair disappears and a probe (letter "E" or "F") appears immediately in the location of one of the two previous stimuli. Youth will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. This paradigm has been modified to facilitate an attention bias away from threat material. In this case, the probe always replaces the neutral stimuli. Thus, although there will be no specific instruction to direct attention away from the threat stimuli, on all trials, the position of the neutral stimulus will indicate the position of the probe.
  Other Names: ABM, attention bias modification, attention training
  Arms: Attention Modification Training
Behavioral: Attention Control Condition — Each trial begins with a fixation cross presented in the center of the computer screen. The cross is then replaced by a face pair presented in the center of the screen. The face pair disappears and a probe (letter "E" or "F") appears immediately in the location of one of the two previous stimuli. Youth will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. This paradigm is not intended to facilitate an attention bias away from threat material. In this case, the probe randomly replaces the threat or neutral stimulus.
  Other Names: ACC
  Arms: Attention Control Training

SUMMARY:
This study aims to test the efficacy and feasibility of administering a computerized attention training program targeting clinical levels of anxiety in Latino youth between the ages of 8-17. 52 youth from Imperial County, a rural and predominantly Latino region, will be randomized to receive either 1) a 12-session attention modification program (AMP) or 2) an attention condition program (non-active treatment). Clinical assessment of symptom severity will be conducted before, during, and after treatment. We hypothesize that at the end of treatment, children who receive the active intervention (AMP) will show (1) decreased attention bias to anxiety-related triggers using an independent measure of attention bias to assess change and (b) reduced anxiety severity. We also hypothesize that this study will be feasible, tolerable, acceptable, and safe in this underserved sample of Latino youth. This study is an initial step towards demonstrating the feasibility of implementing a novel computerized attention training program in anxiety in underserved community samples.

DETAILED DESCRIPTION:
The main aim of this pilot study is to examine the feasibility, tolerability, and acceptability of a computerized attention training program for children who have clinically elevated anxiety. Youth from a rural Latino community, with significant anxiety symptoms (N = 52) will be randomized to an active attention bias modification program (AMP) for four weeks or to an attention control condition (nonactive) for four weeks. Families will be assessed at baseline, mistreatment, post-treatment and 3 month followup. AMP responders will be determined by reduction on a self-report measure of anxiety and a clinician administered assessment. Community health workers (promotoras) will be trained to administer the program to youth. Data will be gathered to examine the feasibility, tolerability, and acceptability of this type of treatment and this mode of service delivery. It is hypothesized that the AMP will be feasible, tolerable, and acceptable to this underserved community sample of ethnic minority youth.

Study Design: Following ascertainment of study eligibility and completion of baseline assessment, youth will be assigned to four weeks of AMP or ACC (attention control condition). All youngsters and their families will undergo a comprehensive baseline assessment and be reassessed at mistreatment, treatment endpoint (week 4) and 3 month followup.

Screening: Youth will be recruited through various mechanisms.

1. Flyers will be posted in primary care clinics in Imperial Valley and Los Angeles County. Clinicas de Salud del Pueblo is a private, non-profit corporation providing primary care services throughout Imperial County. Flyers will be posted in the 10 primary care clinics, located in Imperial County.
2. The second method for recruiting subjects will be through physician referral from providers within the primary care systems. Prior to the study start, all pediatricians/providers will receive information about the study, symptoms of child anxiety, and the use of a short screening measure to assist in detecting child anxiety. If a provider at one of the clinics identifies a child with anxiety or a parent reports that child has symptoms consistent with anxiety (fears, worries, nervousness, unexplained somatic complaints, etc.), the provider will have the option to explain the study to the parent and give them the study brochures. Alternatively, providers, if able, can also ask parents to sign a consent to contact form, giving the research team permission to contact them directly to discuss the study.
3. Providers may also chose to refer the patient to the study promotora who will assist will explaining the study to the participant, screening, and consenting the participants.
4. Flyers will also be posted at Sun Valley Behavioral Medical Center, a private medical clinic that serves the medical and mental health needs of children, adolescents and adults in Imperial County. In this case, parents will be expected to call our research team for more information.
5. The co-PI on this study, Dr. Denise Chavira has an ongoing school based study being conducted with high school students in Imperial Valley. Given that this study covers a range of ages (8-17), we will also recruit from high schools. As part of the existing consent form (for protocol 14-000663), students are asked to check the box if they are interested in participating in future research studies. We will contact those students who have indicated interest in future studies to discuss the current project.

In all of these methods, the community health worker/promotora/e will contact the parent to conduct an initial screen. Thereafter the promotora and/or research coordinator will arrange an in person meeting with the parent and youth to review the consent with the parent and assent form with the youth and administer the eligibility measures. The initial eligibility assessments will not be conducted until all consent/assent forms have been signed and returned to the research team.

At the end of the eligibility visits, the PIs (Chavira and Chang) will review the questionnaires to determine final eligibility. Those who are eligible will process to the baseline visit where they will receive the AMP or ACC program as well as other measures. We have included a table of these measures as well as the assessment schedule in 10.1 section 1.0.

Attention Modification Program: AMP is a modified version of the dot-probe paradigm similar to the original task used by MacLeod, Mathews, and Tata. Each trial begins with a fixation cross presented in the center of the computer screen for 500 ms. The cross is then replaced by a pair of faces presented in the center of the screen for 500 ms. The face pair disappears and a probe (i.e., the letter "E" or "F") appears immediately in the location of one of the two faces. Participants will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. The letter probe will remain on the screen until the participant responds. Response latencies to identify the probe will be recorded from the onset of the presentation of the letter probe to the button press. A total of 288 training trials will be delivered each session. This paradigm has been modified to facilitate an attention bias away from threatening material. In this case, the probe always replaces the neutral face. Thus, although there will be no specific instruction to direct attention away from the threatening face, on all trials, the position of the neutral face will indicate the position of the probe.

Attention Control Condition: Like AMP, the attention control condition is a dot-probe task that begins with a fixation cross presented in the computer screen for 500ms, is followed by a pair of faces (one neutral, one threatening) for 500ms, and then a trial is completed when the face pair disappears and a probe (letter "E" or "F") appears in the location of one of the two faces. Participants will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. The letter probe will remain on the screen until the participant responds. Response latencies to identify the probe will be recorded from the onset of the presentation of the letter probe to the button press. A total of 288 training trials will be delivered each session. However, in this case, the probe replaces both the neutral and threat face 50% of the time.

Assessment. All parents and children enrolled in the study will complete assessments at baseline, mid-treatment, post-treatment and 3 month followup. Assessments will focus on feasibility outcomes and clinical outcome measures. Further, measures of moderating factors will be included in order to better understand variables (e.g., poverty, attention control, acculturation) that may suggest trends in differential treatment response within the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children and parents of children ages 8 through 17 inclusive at the time of initial evaluation 2. Clinically significant levels of anxiety as measured by self-report 3. Unmedicated or on stable medication treatment for at least 6 weeks prior to study entry, with no planned changes for duration of study participation.

  4. Child is fluent English or Spanish speaker, given that all of our assessments as well as the language-based treatment protocol have thus far only been validated in English and Spanish.

  5. Parental Informed Consent and Child Informed Assent. Parents must agree to their child's participation in this protocol. Parents will be asked to fill out self-report questionnaires and participate in assessments that will provide us with more information about their child, however parents are not considered "participants" within this protocol, as all treatment is targeted toward their child.

  6. Child self-identifies as Latino/Hispanic

Exclusion Criteria:

1. Excessive or Problematic Substance Use as reported per initial telephone screening, or significant disruptive behavior problems within the past 3 months.
2. Indication of clinically significant suicidality, mania, or psychotic disorder.
3. Any serious psychiatric, psychosocial, or neurological condition (i.e., ADHD, tourettes, anxiety, severe aggression) requiring immediate treatment.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impression-Severity (CGI-S) and Improvement, (CGI-I) Scales, Pre- to Post-Treatment | through study completion, average of 4 weeks
  Participants receiving a post-treatment CGI-I score of 1 (very much improved) or 2 (much improved) on this one-item, 7-point rating will be considered treatment responders.

SECONDARY OUTCOMES:
Change in Attention Network Task Pre- to Post-Treatment | through study completion, average of 4 weeks
  In this version of the cognitive flanker, participants must indicate whether the central target arrow in a set of 5 arrows is pointing to the left or the right. In congruent trials, all 5 arrows point in the same direction (e.g., →→→→→) while in the incongruent trials, the middle arrow points in the opposite direction as the flanking arrows (e.g., →→←→→). Participants are asked to press the left mouse button if the arrow points to the left and right button if it points to the right.
Change in Visual search task Pre to Post-Treatment | through study completion, average of 4 weeks
  we will include a visual search task as an independent task of attention bias designed to measure spatial attention allocation (Rink, Becker, Kellerman & Roth, 2003). Participants are asked to detect a target stimulus that is embedded in a matrix of distracting stimuli (e.g., a target stimulus, an angry face, might be embedded in a matrix of neutral distractor faces). Attention biases are inferred from faster response times to detect a threatening stimulus in a matrix of neutral stimuli relative to response time to detect neutral stimuli in neutral matrices.
Change in Pediatric Anxiety Rating Scale Pre to Post-treatment | through study completion, average of 4 weeks
  The 50-item PARS is a clinician measure that integrates youth and parent report of the severity of anxiety symptoms, as well as related functional impairment. PARS yields a continuous total score of 0-35.
Change in Screen for Child Anxiety Related Emotional Disorders (SCARED) Pre- to Post-Treatment | through study completion, average of 4 weeks
  The SCARED is a 41-item measure of anxiety symptoms with youth and parent-reported versions, with scores of > 25 indicating significant anxiety (total range 0-82).

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Chang, PhD, Principal Investigator — UCLA Department of Psychiatry; Denise Chavira, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Clinicas de Salud del Pueblo healthcare system, El Centro, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from approximately 52 subjects who are participating in a RCT examining the effectiveness of promotora delivered ABM vs. and active control condition for rural Latino youth with anxiety. The final dataset will include self-reported demographic, clinical symptom, functional impairment, and mental health service use data from questionnaires and interviews with the participants. The dataset will be stripped of identifiers prior to release for sharing. We will make the data and available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. This data will be a part of the NIMH data sharing repository - National Database for Clinical Trials Related to Mental Illness, and made available after study completion.